CLINICAL TRIAL: NCT01011517
Title: Effect of Muscadine Grape Seed Supplementation on Vascular Function in Subjects With or at Risk for Cardiovascular Disease: A Randomized Crossover Trial
Brief Title: Muscadine Grape Seed Supplementation and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB00002611
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Dietary Supplements
Keywords: muscadine grapes; endothelial function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- grape seed supplement (Experimental): Nature's Pearl 650 mg, two capsules daily
  Interventions: Dietary Supplement: Muscadine grape seed supplement
- placebo (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Muscadine grape seed supplement

INTERVENTIONS:
Dietary Supplement: Muscadine grape seed supplement — Nature's Pearl 650 mg, two capsules daily
  Other Names: Nature's Pearl 650 mg, two capsules daily

SUMMARY:
The investigators sought to evaluate the effect of muscadine grape seed supplementation on brachial diameter and flow-mediated vasodilator responses in subjects with, or at risk for cardiovascular disease.

Methods: In a randomized, double-blind, placebo-controlled crossover trial, 50 adults (25 men, 25 women) with one or more cardiac risk factors were randomized to muscadine grape seed (MGS) supplement 1300mg daily vs.. placebo for 4 weeks each, with a 4-week washout between study periods. Resting diameter and endothelial function measured using brachial flow-mediated dilation (FMD) were determined at the beginning and end of each study period.

DETAILED DESCRIPTION:
Study Participants Participants were adult male and non-pregnant female outpatients ages 18-65 with one or more of the following cardiovascular risk factors: hypertension (blood pressure ≥ 140/90 or current treatment for hypertension); dyslipidemia (total cholesterol > 220 mg/dL + LDL cholesterol > 130 mg/dL, or current use of lipid-lowering medications); or controlled type 2 diabetes mellitus (glycated hemoglobin < 8.0 % with or without medication). Subjects with a history of coronary artery disease (any history of myocardial infarction or coronary revascularization) were also eligible for participation. Subjects were excluded if they had a history of congestive heart failure (any classification), unstable angina or acute coronary syndrome within the last 30 days, uncontrolled hypertension (blood pressure ≥ 170/100 mm/Hg), type 1 diabetes mellitus, uncontrolled type 2 diabetes mellitus (HbA1C ≥ 8.0%), history of gastrointestinal disease or surgery affecting absorption, peripheral arterial disease, diagnosis of active cancer (excluding squamous cell or basal cell skin cancer), current use of long-acting nitrate compounds such as isosorbide dinitrate or nitroglycerin, recent change in any medications (last 30 days), active plan to change diet or exercise patterns, history of hypersensitivity to any compound in the intervention or placebo, or history of intolerance to nitrates.

Study Design The study was a double-blind, randomized crossover design to evaluate the effects of muscadine grape seed supplementation (Nature's Pearl 650 mg, two capsules daily.) The phytochemical profile of the supplement is presented in Table 1. The trial consisted of a screening visit followed by baseline and closeout visits for two study treatment periods (4 weeks each), separated by a 4-week washout period (total of 5 visits over 14 weeks).Endothelial function was assessed at the beginning and end of each study period using brachial artery flow-mediated dilation (brachial FMD - described below). A fasting blood sample was obtained at the open and close of each study period for measurement of lipids, inflammatory markers, and markers of antioxidant capacity and oxidative stress. Participants were asked to abstain from red wine, antioxidant vitamin supplements (including vitamin E, vitamin C, and beta-carotene supplements, more than 1 cup of black or green tea daily, and other grape seed supplements. Multivitamin supplements were permitted as long as they were taken for the study duration.

Endothelial Function Study Protocol Details for the brachial FMD protocol, automated analysis and reproducibility have been published previously {Herrington 2001}. Briefly, subjects rested in a quiet, temperature-controlled room for 15 minutes. A standard (pediatric) cuff was placed on the right forearm 2 inches (5 cm) below the antecubital fossa. Once the transducer position was established over the left brachial artery, continuous scanning of the brachial artery was obtained for 2 minutes before the cuff occlusion, 4 minutes of cuff occlusion, and 2 minutes immediately after cuff release. Data were analyzed with an automated analysis system that determines changes in brachial artery diameter for 2 minutes after cuff release.

Statistical Analysis The effects of supplementation with muscadine grape seeds and placebo were compared using paired t-tests and mixed linear models to take into account treatment order and period effects. The mixed linear models were also used to formally test for a residual effect of treatment in those subjects receiving active treatment in the first treatment period. Stratified analyses were performed to look for evidence of differential effects by age, gender, prevalent heart disease or heart disease risk factors. Nominal 2-tailed p-values are presented for the primary outcome (percent change in brachial diameter) and for all secondary outcomes. All analyses were performed using SAS v. 9.1 (Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

* adult male and non-pregnant female outpatients, with
* hypertension (blood pressure ≥ 140/90 or current treatment for hypertension), or
* dyslipidemia (total cholesterol > 220 mg/dL + LDL cholesterol > 130 mg/dL, or current use of lipid-lowering medications), or
* controlled type 2 diabetes mellitus (glycated hemoglobin < 8.0 % with or without medication).

Exclusion Criteria:

* history of congestive heart failure (any classification)
* unstable angina or acute coronary syndrome within the last 30 days,
* uncontrolled hypertension (blood pressure ≥ 170/100 mm/Hg),
* type 1 diabetes mellitus,
* uncontrolled type 2 diabetes mellitus (HbA1C ≥ 8.0%),
* history of gastrointestinal disease or surgery affecting absorption,
* peripheral arterial disease,
* diagnosis of active cancer (excluding squamous cell or basal cell skin cancer),
* current use of long-acting nitrate compounds such as isosorbide dinitrate or nitroglycerin,
* recent change in any medications (last 30 days),
* active plan to change diet or exercise patterns,
* history of hypersensitivity to any compound in the intervention or placebo,
* history of intolerance to nitrates

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Brachial Artery Flow mediated dilation | 1 month

SECONDARY OUTCOMES:
Plasma markers of inflammation and anitoxidant capacity | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: David Herrington, MD, MHS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States